CLINICAL TRIAL: NCT07175051
Title: Targeting the Pathophysiology of Sickle Cell-Related Kidney Disease Using the SGLT2 Inhibitors, Empagliflozin
Acronym: EMPA-CKD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Santosh L Saraf, Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0637
Record Dates: First submitted 2025-08-21; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Anemia (HbSS, or HbSβ-thalassemia0); Albuminuria
Keywords: Empa-CKD; Sickle Cell-Related Kidney Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Albuminuria | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Empagliflozin
  Interventions: Drug: Empagliflozin (oral)

INTERVENTIONS:
Drug: Empagliflozin (oral) — 10 mg

SUMMARY:
Sickle cell anemia (SCA) is an inherited red blood disorder. The kidneys are among the most commonly affected organ systems in SCA. The Food and Drug Administration (FDA) has approved empagliflozin as a treatment to reduce the decline of kidney function in those with kidney disease. The proposed research study aims to determine whether empagliflozin can prevent the progression of kidney dysfunction in patients with sickle cell anemia (SCA) who are at high risk of developing advanced chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Documentation of SCA genotype (HbSS or HbSβ0-thalassemia)
* Albuminuria defined by a UACR of 100 - 2,000 mg/g creatinine at the screening
* Hemoglobin (Hb) ≥ 5.5 g/dL during screening
* For participants taking Endari, the dose of Endari must be stable for at least one month prior to signing the ICF and with no anticipated need for dose adjustments during the study
* For participants on crizanlizumab or chronic red blood cell transfusions, the therapy must have started at least 3 months prior to consent
* For participants taking an angiotensin converting enzyme inhibitor (ACEi) or angiotensin II receptor blocker (ARB), the dose must be stable for at least 3 months prior to signing the ICF and with no anticipated need for dose adjustments during the study, in the opinion of the Investigator
* Participants must demonstrate regular compliance with clinic visits and outpatient management
* Participants, if female and of childbearing potential, will use highly effective methods of contraception from study start to 30 days after the last dose of the study drug
* Participant has provided documented informed consent or assent

Exclusion Criteria:

* Concurrent diagnosis of diabetes mellitus
* Female who is breast feeding, pregnant, or unwilling to use birth control as described in the protocol
* Prior hypersensitivity or intolerance to a sodium-glucose cotransporter-2 inhibitor (SGLT2i)
* Active or open leg ankle ulcer
* Chronic urinary tract infection
* Hospitalized for sickle cell crisis or other vaso-occlusive event within 14 days prior to signing consent
* Hepatic dysfunction characterized by alanine aminotransferase (ALT) >5× ULN
* Participants with acute bacterial infection requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed
* Participants with known active hepatitis A, B, or C or who are known to be human immunodeficiency virus (HIV) positive
* Moderate to severe CKD (defined by an eGFR < 30 mL/min/1.73m2, on chronic dialysis, or having received a kidney transplantation)
* History of malignancy within the past 2 years prior to treatment Day 1 requiring chemotherapy and/or radiation (with the exception of local therapy for non-melanoma skin malignancy)
* History of unstable or deteriorating cardiac or pulmonary disease within 6 months prior to consent including but not limited to the following:

  1. Unstable angina pectoris or myocardial infarction or elective coronary intervention
  2. Uncontrolled clinically significant arrhythmias
* Any condition affecting drug absorption, such as major surgery involving the stomach (e.g. bariatric surgery) or small intestine (prior cholecystectomy is acceptable)
* Participated in another clinical trial of an investigational agent (or medical device) within 30 days or 5 half-lives of agent, whichever is longer, or is currently participating in another trial of an investigational agent or medical device)
* Medical, psychological, or behavioral conditions, which, in the opinion of the Investigator, may preclude safe participation, confound study interpretation, interfere with compliance, or preclude informed consent
* Contraindication to MRI (certain pacemakers, electronic implants, shrapnel in the eyes, or certain intracranial aneurysm clips)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of empagliflozin - urine biomarker: Adenosine | From enrollment to the end of treatment at 48 weeks
  Adenosine (umol/g creatinine) average values from Screening & Visit 1 compared to average values from Visit 5 & 6.
Efficacy of empagliflozin - urine biomarker: Nephrin | From enrollment to the end of treatment at 48 weeks
  Nephrin (ng/g creatinine) average values from Screening & Visit 1 compared to average values from Visit 5 & 6.
Efficacy of empagliflozin - urine biomarker: Kidney injury molecule-1 | From enrollment to the end of treatment at 48 weeks
  Kidney injury molecule-1 (ng/g creatinine) average values from Screening & Visit 1 compared to average values from Visit 5 & 6.
Efficacy of empagliflozin R2* Cortical Oxygenation on kidney fMRI | From enrollment to the end of treatment at 48 weeks
  fMRI-derived R2* average values from Visit 1 compared to the values from Visit 6.

SECONDARY OUTCOMES:
Effects of empagliflozin on UACR | From enrollment to the end of treatment at 48 weeks
  Change in UACR (mg/g creatinine) average values from Screening & Visit 1 compared to average values from Visit 5 & 6
Effects of empagliflozin on 24-hour urine protein | From enrollment to the end of treatment at 48 weeks
  24-hour urine protein (g/24 hours) average values from Screening & Visit 1 compared to average values from Visit 5 & 6.
Effects of empagliflozin on measures of eGFR | From enrollment to the end of treatment at 48 weeks
  eGFR calculated by race-free serum creatinine and cystatin C-based equations (mL/min/1.73m2), average values from Screening & Visit 1 compared to average values from Visit 5 & 6
Effects of empagliflozin on serum biomarker: suPAR | From enrollment to the end of treatment at 48 weeks
  suPAR pg/mL average values from Screening & Visit 1 compared to average values from Visit 5 & 6.
Effects of empagliflozin on serum biomarker: Et-1 | From enrollment to the end of treatment at 48 weeks
  ET-1 pg/mL average values from Screening & Visit 1 compared to average values from Visit 5 & 6.
Effects of empagliflozin on serum biomarker: VCAM-1 | From enrollment to the end of treatment at 48 weeks
  VCAM-1 ng/mL average values from Screening & Visit 1 compared to average values from Visit 5 & 6.
Effects of empagliflozin on serum biomarker: sFLTI-1 | From enrollment to the end of treatment at 48 weeks
  sFLTI-1 ng/L average values from Screening & Visit 1 compared to average values from Visit 5 & 6.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Sickle Cell Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srivastava A, Cai X, Lee J, Li W, Larive B, Kendrick C, Gassman JJ, Middleton JP, Carr J, Raphael KL, Cheung AK, Raj DS, Chonchol MB, Fried LF, Block GA, Sprague SM, Wolf M, Ix JH, Prasad PV, Isakova T. Kidney Functional Magnetic Resonance Imaging and Change in eGFR in Individuals with CKD. Clin J Am Soc Nephrol. 2020 Jun 8;15(6):776-783. doi: 10.2215/CJN.13201019. Epub 2020 Apr 28. PMID 32345747
- [Background] Prasad PV, Li LP, Thacker JM, Li W, Hack B, Kohn O, Sprague SM. Cortical Perfusion and Tubular Function as Evaluated by Magnetic Resonance Imaging Correlates with Annual Loss in Renal Function in Moderate Chronic Kidney Disease. Am J Nephrol. 2019;49(2):114-124. doi: 10.1159/000496161. Epub 2019 Jan 22. PMID 30669143
- [Background] Prasad PV, Li W, Raj DS, Carr J, Carr M, Thacker J, Li LP, Wang C, Sprague SM, Ix JH, Chonchol M, Block G, Cheung AK, Raphael K, Gassman J, Wolf M, Fried LF, Isakova T; CKD Optimal Management with BInders and NicotinamidE (COMBINE) study group. Multicenter Study Evaluating Intrarenal Oxygenation and Fibrosis Using Magnetic Resonance Imaging in Individuals With Advanced CKD. Kidney Int Rep. 2018 Jul 7;3(6):1467-1472. doi: 10.1016/j.ekir.2018.07.006. eCollection 2018 Nov. No abstract available. PMID 30450473
- [Background] Wang J, Silaghi P, Guo C, Harro D, Eitzman DT. Inhibition of sodium-glucose cotransporter-2 improves anaemia in mice and humans with sickle cell disease, and reduces infarct size in a murine stroke model. J Cell Mol Med. 2024 Sep;28(17):e70091. doi: 10.1111/jcmm.70091. PMID 39267208
- [Background] Tian Q, Guo K, Deng J, Zhong Y, Yang L. Effects of SGLT2 inhibitors on haematocrit and haemoglobin levels and the associated cardiorenal benefits in T2DM patients: A meta-analysis. J Cell Mol Med. 2022 Jan;26(2):540-547. doi: 10.1111/jcmm.17115. Epub 2021 Dec 8. PMID 34878225
- [Background] von Eynatten M, Baumann M, Heemann U, Zdunek D, Hess G, Nawroth PP, Bierhaus A, Humpert PM. Urinary L-FABP and anaemia: distinct roles of urinary markers in type 2 diabetes. Eur J Clin Invest. 2010 Feb;40(2):95-102. doi: 10.1111/j.1365-2362.2009.02220.x. Epub 2009 Nov 11. PMID 19912308
- [Background] Johannes T, Mik EG, Nohe B, Unertl KE, Ince C. Acute decrease in renal microvascular PO2 during acute normovolemic hemodilution. Am J Physiol Renal Physiol. 2007 Feb;292(2):F796-803. doi: 10.1152/ajprenal.00206.2006. Epub 2006 Oct 31. PMID 17077389
- [Background] Grune T, Sommerburg O, Siems WG. Oxidative stress in anemia. Clin Nephrol. 2000 Feb;53(1 Suppl):S18-22. PMID 10746801
- [Background] Asnani MR, Lynch O, Reid ME. Determining glomerular filtration rate in homozygous sickle cell disease: utility of serum creatinine based estimating equations. PLoS One. 2013 Jul 19;8(7):e69922. doi: 10.1371/journal.pone.0069922. Print 2013. PMID 23894560
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Thrower A, Ciccone EJ, Maitra P, Derebail VK, Cai J, Ataga KI. Effect of renin-angiotensin-aldosterone system blocking agents on progression of glomerulopathy in sickle cell disease. Br J Haematol. 2019 Jan;184(2):246-252. doi: 10.1111/bjh.15651. Epub 2018 Nov 21. PMID 30460977
- [Background] Wright JT Jr, Bakris G, Greene T, Agodoa LY, Appel LJ, Charleston J, Cheek D, Douglas-Baltimore JG, Gassman J, Glassock R, Hebert L, Jamerson K, Lewis J, Phillips RA, Toto RD, Middleton JP, Rostand SG; African American Study of Kidney Disease and Hypertension Study Group. Effect of blood pressure lowering and antihypertensive drug class on progression of hypertensive kidney disease: results from the AASK trial. JAMA. 2002 Nov 20;288(19):2421-31. doi: 10.1001/jama.288.19.2421. PMID 12435255
- [Background] Heerspink HJ, Kropelin TF, Hoekman J, de Zeeuw D; Reducing Albuminuria as Surrogate Endpoint (REASSURE) Consortium. Drug-Induced Reduction in Albuminuria Is Associated with Subsequent Renoprotection: A Meta-Analysis. J Am Soc Nephrol. 2015 Aug;26(8):2055-64. doi: 10.1681/ASN.2014070688. Epub 2014 Nov 24. PMID 25421558
- [Background] Abo-Zenah H, Moharram M, El Nahas AM. Cardiorenal risk prevalence in sickle cell hemoglobinopathy. Nephron Clin Pract. 2009;112(2):c98-c106. doi: 10.1159/000213897. Epub 2009 Apr 23. PMID 19390209
- [Background] Mayr A, Pfeifer F. The characterization of the nv-gvpACNOFGH gene cluster involved in gas vesicle formation in Natronobacterium vacuolatum. Arch Microbiol. 1997 Jul;168(1):24-32. doi: 10.1007/s002030050465. PMID 9211710
- [Background] Roscioni SS, Lambers Heerspink HJ, de Zeeuw D. Microalbuminuria: target for renoprotective therapy PRO. Kidney Int. 2014 Jul;86(1):40-9. doi: 10.1038/ki.2013.490. Epub 2014 Apr 23. PMID 24759154
- [Background] Lambers Heerspink HJ, Gansevoort RT. Albuminuria Is an Appropriate Therapeutic Target in Patients with CKD: The Pro View. Clin J Am Soc Nephrol. 2015 Jun 5;10(6):1079-88. doi: 10.2215/CJN.11511114. Epub 2015 Apr 17. PMID 25887073
- [Background] Lee MMY, Gillis KA, Brooksbank KJM, Allwood-Spiers S, Hall Barrientos P, Wetherall K, Roditi G, AlHummiany B, Berry C, Campbell RT, Chong V, Coyle L, Docherty KF, Dreisbach JG, Kuehn B, Labinjoh C, Lang NN, Lennie V, Mangion K, McConnachie A, Murphy CL, Petrie CJ, Petrie JR, Sharma K, Sourbron S, Speirits IA, Thompson J, Welsh P, Woodward R, Wright A, Radjenovic A, McMurray JJV, Jhund PS, Petrie MC, Sattar N, Mark PB. Effect of Empagliflozin on Kidney Biochemical and Imaging Outcomes in Patients With Type 2 Diabetes, or Prediabetes, and Heart Failure with Reduced Ejection Fraction (SUGAR-DM-HF). Circulation. 2022 Jul 26;146(4):364-367. doi: 10.1161/CIRCULATIONAHA.122.059851. Epub 2022 Jul 25. No abstract available. PMID 35877829
- [Background] Zanchi A, Burnier M, Muller ME, Ghajarzadeh-Wurzner A, Maillard M, Loncle N, Milani B, Dufour N, Bonny O, Pruijm M. Acute and Chronic Effects of SGLT2 Inhibitor Empagliflozin on Renal Oxygenation and Blood Pressure Control in Nondiabetic Normotensive Subjects: A Randomized, Placebo-Controlled Trial. J Am Heart Assoc. 2020 Jul 7;9(13):e016173. doi: 10.1161/JAHA.119.016173. Epub 2020 Jun 20. PMID 32567439
- [Background] Ritt M, Janka R, Schneider MP, Martirosian P, Hornegger J, Bautz W, Uder M, Schmieder RE. Measurement of kidney perfusion by magnetic resonance imaging: comparison of MRI with arterial spin labeling to para-aminohippuric acid plasma clearance in male subjects with metabolic syndrome. Nephrol Dial Transplant. 2010 Apr;25(4):1126-33. doi: 10.1093/ndt/gfp639. Epub 2009 Nov 24. PMID 19934080
- [Background] Prasad PV, Kim D, Kaiser AM, Chavez D, Gladstone S, Li W, Buxton RB, Edelman RR. Noninvasive comprehensive characterization of renal artery stenosis by combination of STAR angiography and EPISTAR perfusion imaging. Magn Reson Med. 1997 Nov;38(5):776-87. doi: 10.1002/mrm.1910380514. PMID 9358452
- [Background] Martirosian P, Klose U, Mader I, Schick F. FAIR true-FISP perfusion imaging of the kidneys. Magn Reson Med. 2004 Feb;51(2):353-61. doi: 10.1002/mrm.10709. PMID 14755661
- [Background] Prasad PV. Evaluation of intra-renal oxygenation by BOLD MRI. Nephron Clin Pract. 2006;103(2):c58-65. doi: 10.1159/000090610. Epub 2006 Mar 10. PMID 16543757
- [Background] Prasad PV, Edelman RR, Epstein FH. Noninvasive evaluation of intrarenal oxygenation with BOLD MRI. Circulation. 1996 Dec 15;94(12):3271-5. doi: 10.1161/01.cir.94.12.3271. PMID 8989140
- [Background] Li LP, Halter S, Prasad PV. Blood oxygen level-dependent MR imaging of the kidneys. Magn Reson Imaging Clin N Am. 2008 Nov;16(4):613-25, viii. doi: 10.1016/j.mric.2008.07.008. PMID 18926426
- [Background] Berchtold L, Friedli I, Crowe LA, Martinez C, Moll S, Hadaya K, de Perrot T, Combescure C, Martin PY, Vallee JP, de Seigneux S. Validation of the corticomedullary difference in magnetic resonance imaging-derived apparent diffusion coefficient for kidney fibrosis detection: a cross-sectional study. Nephrol Dial Transplant. 2020 Jun 1;35(6):937-945. doi: 10.1093/ndt/gfy389. PMID 30608554
- [Background] Inoue T, Kozawa E, Okada H, Inukai K, Watanabe S, Kikuta T, Watanabe Y, Takenaka T, Katayama S, Tanaka J, Suzuki H. Noninvasive evaluation of kidney hypoxia and fibrosis using magnetic resonance imaging. J Am Soc Nephrol. 2011 Aug;22(8):1429-34. doi: 10.1681/ASN.2010111143. Epub 2011 Jul 14. PMID 21757771
- [Background] Wang W, Yu Y, Wen J, Zhang M, Chen J, Cheng D, Zhang L, Liu Z. Combination of Functional Magnetic Resonance Imaging and Histopathologic Analysis to Evaluate Interstitial Fibrosis in Kidney Allografts. Clin J Am Soc Nephrol. 2019 Sep 6;14(9):1372-1380. doi: 10.2215/CJN.00020119. Epub 2019 Aug 15. PMID 31416890
- [Background] Mao W, Zhou J, Zeng M, Ding Y, Qu L, Chen C, Ding X, Wang Y, Fu C, Gu F. Intravoxel incoherent motion diffusion-weighted imaging for the assessment of renal fibrosis of chronic kidney disease: A preliminary study. Magn Reson Imaging. 2018 Apr;47:118-124. doi: 10.1016/j.mri.2017.12.010. Epub 2017 Dec 5. PMID 29217491
- [Background] Togao O, Doi S, Kuro-o M, Masaki T, Yorioka N, Takahashi M. Assessment of renal fibrosis with diffusion-weighted MR imaging: study with murine model of unilateral ureteral obstruction. Radiology. 2010 Jun;255(3):772-80. doi: 10.1148/radiol.10091735. Epub 2010 Apr 20. PMID 20406881
- [Background] Le Bihan D, Breton E, Lallemand D, Aubin ML, Vignaud J, Laval-Jeantet M. Separation of diffusion and perfusion in intravoxel incoherent motion MR imaging. Radiology. 1988 Aug;168(2):497-505. doi: 10.1148/radiology.168.2.3393671.
- [Background] Odudu A, Nery F, Harteveld AA, Evans RG, Pendse D, Buchanan CE, Francis ST, Fernandez-Seara MA. Arterial spin labelling MRI to measure renal perfusion: a systematic review and statement paper. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii15-ii21. doi: 10.1093/ndt/gfy180. PMID 30137581
- [Background] Caroli A, Schneider M, Friedli I, Ljimani A, De Seigneux S, Boor P, Gullapudi L, Kazmi I, Mendichovszky IA, Notohamiprodjo M, Selby NM, Thoeny HC, Grenier N, Vallee JP. Diffusion-weighted magnetic resonance imaging to assess diffuse renal pathology: a systematic review and statement paper. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii29-ii40. doi: 10.1093/ndt/gfy163. PMID 30137580
- [Background] Pruijm M, Mendichovszky IA, Liss P, Van der Niepen P, Textor SC, Lerman LO, Krediet CTP, Caroli A, Burnier M, Prasad PV. Renal blood oxygenation level-dependent magnetic resonance imaging to measure renal tissue oxygenation: a statement paper and systematic review. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii22-ii28. doi: 10.1093/ndt/gfy243. PMID 30137579
- [Background] Selby NM, Blankestijn PJ, Boor P, Combe C, Eckardt KU, Eikefjord E, Garcia-Fernandez N, Golay X, Gordon I, Grenier N, Hockings PD, Jensen JD, Joles JA, Kalra PA, Kramer BK, Mark PB, Mendichovszky IA, Nikolic O, Odudu A, Ong ACM, Ortiz A, Pruijm M, Remuzzi G, Rorvik J, de Seigneux S, Simms RJ, Slatinska J, Summers P, Taal MW, Thoeny HC, Vallee JP, Wolf M, Caroli A, Sourbron S. Magnetic resonance imaging biomarkers for chronic kidney disease: a position paper from the European Cooperation in Science and Technology Action PARENCHIMA. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii4-ii14. doi: 10.1093/ndt/gfy152. PMID 30137584
- [Background] Lebensburger JD, Gossett J, Zahr R, Wang WC, Ataga KI, Estepp JH, Kang G, Hankins JS. High bias and low precision for estimated versus measured glomerular filtration rate in pediatric sickle cell anemia. Haematologica. 2021 Jan 1;106(1):295-298. doi: 10.3324/haematol.2019.242156. No abstract available. PMID 32107332
- [Background] Zahr RS, Yee ME, Weaver J, Twombley K, Matar RB, Aviles D, Sreedharan R, Rheault MN, Malatesta-Muncher R, Stone H, Srivastava T, Kapur G, Baddi P, Volovelsky O, Pelletier J, Gbadegesin R, Seeherunvong W, Patel HP, Greenbaum LA. Kidney biopsy findings in children with sickle cell disease: a Midwest Pediatric Nephrology Consortium study. Pediatr Nephrol. 2019 Aug;34(8):1435-1445. doi: 10.1007/s00467-019-04237-3. Epub 2019 Apr 3. PMID 30945006
- [Background] Sun R, Srivastava A, Derebail VK, Han J, Molokie RE, Gordeuk V, Saraf SL. GLP-1 agonists and SGLT-2 inhibitors in adults with sickle cell disease. Am J Hematol. 2024 Aug;99(8):1610-1612. doi: 10.1002/ajh.27348. Epub 2024 Apr 24. No abstract available. PMID 38655752
- [Background] Brenner BM, Cooper ME, de Zeeuw D, Keane WF, Mitch WE, Parving HH, Remuzzi G, Snapinn SM, Zhang Z, Shahinfar S; RENAAL Study Investigators. Effects of losartan on renal and cardiovascular outcomes in patients with type 2 diabetes and nephropathy. N Engl J Med. 2001 Sep 20;345(12):861-9. doi: 10.1056/NEJMoa011161. PMID 11565518
- [Background] Randomised placebo-controlled trial of effect of ramipril on decline in glomerular filtration rate and risk of terminal renal failure in proteinuric, non-diabetic nephropathy. The GISEN Group (Gruppo Italiano di Studi Epidemiologici in Nefrologia). Lancet. 1997 Jun 28;349(9069):1857-63. PMID 9217756
- [Background] de Zeeuw D, Remuzzi G, Parving HH, Keane WF, Zhang Z, Shahinfar S, Snapinn S, Cooper ME, Mitch WE, Brenner BM. Albuminuria, a therapeutic target for cardiovascular protection in type 2 diabetic patients with nephropathy. Circulation. 2004 Aug 24;110(8):921-7. doi: 10.1161/01.CIR.0000139860.33974.28. Epub 2004 Aug 9. PMID 15302780
- [Background] Cherney DZI, Zinman B, Inzucchi SE, Koitka-Weber A, Mattheus M, von Eynatten M, Wanner C. Effects of empagliflozin on the urinary albumin-to-creatinine ratio in patients with type 2 diabetes and established cardiovascular disease: an exploratory analysis from the EMPA-REG OUTCOME randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2017 Aug;5(8):610-621. doi: 10.1016/S2213-8587(17)30182-1. Epub 2017 Jun 27. PMID 28666775
- [Background] Ferreira JP, Zannad F, Butler J, Filippatos G, Pocock SJ, Brueckmann M, Steubl D, Schueler E, Anker SD, Packer M. Association of Empagliflozin Treatment With Albuminuria Levels in Patients With Heart Failure: A Secondary Analysis of EMPEROR-Pooled. JAMA Cardiol. 2022 Nov 1;7(11):1148-1159. doi: 10.1001/jamacardio.2022.2924. PMID 36129693
- [Background] Saraf SL, Han J, Ruiz MA, et al. Defining and Predicting Rapid Egfr Decline in Sickle Cell Disease. Blood. 2021;138.
- [Background] Schaub JA, AlAkwaa FM, McCown PJ, Naik AS, Nair V, Eddy S, Menon R, Otto EA, Demeke D, Hartman J, Fermin D, O'Connor CL, Subramanian L, Bitzer M, Harned R, Ladd P, Pyle L, Pennathur S, Inoki K, Hodgin JB, Brosius FC 3rd, Nelson RG, Kretzler M, Bjornstad P. SGLT2 inhibitors mitigate kidney tubular metabolic and mTORC1 perturbations in youth-onset type 2 diabetes. J Clin Invest. 2023 Mar 1;133(5):e164486. doi: 10.1172/JCI164486. PMID 36637914
- [Background] Wang J, Tran J, Wang H, Guo C, Harro D, Campbell AD, Eitzman DT. mTOR Inhibition improves anaemia and reduces organ damage in a murine model of sickle cell disease. Br J Haematol. 2016 Aug;174(3):461-9. doi: 10.1111/bjh.14057. Epub 2016 Mar 31. PMID 27030515
- [Background] Bilan VP, Schneider F, Novelli EM, Kelley EE, Shiva S, Gladwin MT, Jackson EK, Tofovic SP. Experimental intravascular hemolysis induces hemodynamic and pathological pulmonary hypertension: association with accelerated purine metabolism. Pulm Circ. 2018 Jul-Sep;8(3):2045894018791557. doi: 10.1177/2045894018791557. Epub 2018 Jul 13. PMID 30003836
- [Background] Gurkan S, Scarponi KJ, Hotchkiss H, Savage B, Drachtman R. Lactate dehydrogenase as a predictor of kidney involvement in patients with sickle cell anemia. Pediatr Nephrol. 2010 Oct;25(10):2123-7. doi: 10.1007/s00467-010-1560-8. Epub 2010 Jun 2. PMID 20517617
- [Background] Maier-Redelsperger M, Levy P, Lionnet F, Stankovic K, Haymann JP, Lefevre G, Avellino V, Perol JP, Girot R, Elion J. Strong association between a new marker of hemolysis and glomerulopathy in sickle cell anemia. Blood Cells Mol Dis. 2010 Dec 15;45(4):289-92. doi: 10.1016/j.bcmd.2010.08.001. Epub 2010 Sep 15. PMID 20833087
- [Background] Nuffield Department of Population Health Renal Studies Group; SGLT2 inhibitor Meta-Analysis Cardio-Renal Trialists' Consortium. Impact of diabetes on the effects of sodium glucose co-transporter-2 inhibitors on kidney outcomes: collaborative meta-analysis of large placebo-controlled trials. Lancet. 2022 Nov 19;400(10365):1788-1801. doi: 10.1016/S0140-6736(22)02074-8. Epub 2022 Nov 6. PMID 36351458
- [Background] The EMPA-KIDNEY Collaborative Group; Herrington WG, Staplin N, Wanner C, Green JB, Hauske SJ, Emberson JR, Preiss D, Judge P, Mayne KJ, Ng SYA, Sammons E, Zhu D, Hill M, Stevens W, Wallendszus K, Brenner S, Cheung AK, Liu ZH, Li J, Hooi LS, Liu W, Kadowaki T, Nangaku M, Levin A, Cherney D, Maggioni AP, Pontremoli R, Deo R, Goto S, Rossello X, Tuttle KR, Steubl D, Petrini M, Massey D, Eilbracht J, Brueckmann M, Landray MJ, Baigent C, Haynes R. Empagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2023 Jan 12;388(2):117-127. doi: 10.1056/NEJMoa2204233. Epub 2022 Nov 4. PMID 36331190
- [Background] Heerspink HJL, Jongs N, Chertow GM, Langkilde AM, McMurray JJV, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Greene T; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on the rate of decline in kidney function in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):743-754. doi: 10.1016/S2213-8587(21)00242-4. Epub 2021 Oct 4. PMID 34619108
- [Background] Jongs N, Greene T, Chertow GM, McMurray JJV, Langkilde AM, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on urinary albumin excretion in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):755-766. doi: 10.1016/S2213-8587(21)00243-6. Epub 2021 Oct 4. PMID 34619106
- [Background] Sylvester RD, Khong TK. Dapagliflozin in people with chronic kidney disease. Drug Ther Bull. 2023 Aug;61(8):118-119. doi: 10.1136/dtb.2023.000022. Epub 2023 May 31. PMID 37257897
- [Background] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Background] Kogot-Levin A, Hinden L, Riahi Y, Israeli T, Tirosh B, Cerasi E, Mizrachi EB, Tam J, Mosenzon O, Leibowitz G. Proximal Tubule mTORC1 Is a Central Player in the Pathophysiology of Diabetic Nephropathy and Its Correction by SGLT2 Inhibitors. Cell Rep. 2020 Jul 28;32(4):107954. doi: 10.1016/j.celrep.2020.107954. PMID 32726619
- [Background] Deleyto-Seldas N, Efeyan A. The mTOR-Autophagy Axis and the Control of Metabolism. Front Cell Dev Biol. 2021 Jul 1;9:655731. doi: 10.3389/fcell.2021.655731. eCollection 2021. PMID 34277603
- [Background] Tuttle KR. Digging deep into cells to find mechanisms of kidney protection by SGLT2 inhibitors. J Clin Invest. 2023 Mar 1;133(5):e167700. doi: 10.1172/JCI167700. PMID 36856116
- [Background] Thomson SC, Rieg T, Miracle C, Mansoury H, Whaley J, Vallon V, Singh P. Acute and chronic effects of SGLT2 blockade on glomerular and tubular function in the early diabetic rat. Am J Physiol Regul Integr Comp Physiol. 2012 Jan 1;302(1):R75-83. doi: 10.1152/ajpregu.00357.2011. Epub 2011 Sep 21. PMID 21940401
- [Background] Upadhyay A. SGLT2 Inhibitors and Kidney Protection: Mechanisms Beyond Tubuloglomerular Feedback. Kidney360. 2024 May 1;5(5):771-782. doi: 10.34067/KID.0000000000000425. Epub 2024 Mar 25. PMID 38523127
- [Background] Foucan L, Bourhis V, Bangou J, Merault L, Etienne-Julan M, Salmi RL. A randomized trial of captopril for microalbuminuria in normotensive adults with sickle cell anemia. Am J Med. 1998 Apr;104(4):339-42. doi: 10.1016/s0002-9343(98)00056-4. PMID 9576406
- [Background] Yee ME, Lane PA, Archer DR, Joiner CH, Eckman JR, Guasch A. Losartan therapy decreases albuminuria with stable glomerular filtration and permselectivity in sickle cell anemia. Blood Cells Mol Dis. 2018 Mar;69:65-70. doi: 10.1016/j.bcmd.2017.09.006. Epub 2017 Sep 21. PMID 28951038
- [Background] Quinn CT, Saraf SL, Gordeuk VR, Fitzhugh CD, Creary SE, Bodas P, George A, Raj AB, Nero AC, Terrell CE, McCord L, Lane A, Ackerman HC, Yang Y, Niss O, Taylor MD, Devarajan P, Malik P. Losartan for the nephropathy of sickle cell anemia: A phase-2, multicenter trial. Am J Hematol. 2017 Sep;92(9):E520-E528. doi: 10.1002/ajh.24810. Epub 2017 Jul 19. PMID 28589652
- [Background] Saraf SL, Zhang X, Shah B, Kanias T, Gudehithlu KP, Kittles R, Machado RF, Arruda JA, Gladwin MT, Singh AK, Gordeuk VR. Genetic variants and cell-free hemoglobin processing in sickle cell nephropathy. Haematologica. 2015 Oct;100(10):1275-84. doi: 10.3324/haematol.2015.124875. Epub 2015 Jul 23. PMID 26206798
- [Background] Ren G, Setty S, Zhang X, Susma A, Ruiz MA, Minshall RD, Lash JP, Gordeuk VR, Saraf SL. Improvement of hemolytic anemia with GBT1118 is renoprotective in transgenic sickle mice. Blood Adv. 2022 Aug 9;6(15):4403-4407. doi: 10.1182/bloodadvances.2022007809. PMID 35759756
- [Background] Gladwin MT, Kanias T, Kim-Shapiro DB. Hemolysis and cell-free hemoglobin drive an intrinsic mechanism for human disease. J Clin Invest. 2012 Apr;122(4):1205-8. doi: 10.1172/JCI62972. Epub 2012 Mar 26. PMID 22446184
- [Background] Kasztan M, Fox BM, Lebensburger JD, Hyndman KA, Speed JS, Pollock JS, Pollock DM. Hyperfiltration predicts long-term renal outcomes in humanized sickle cell mice. Blood Adv. 2019 May 14;3(9):1460-1475. doi: 10.1182/bloodadvances.2018028878. PMID 31064747
- [Background] Belisario AR, de Almeida JA, Mendes FG, da Silva DMM, Planes W, Rezende PV, Silva CM, Brito AC, Sales RR, Viana MB, Simoes E Silva AC. Prevalence and risk factors for albuminuria and glomerular hyperfiltration in a large cohort of children with sickle cell anemia. Am J Hematol. 2020 May;95(5):E125-E128. doi: 10.1002/ajh.25763. Epub 2020 Feb 29. No abstract available. PMID 32083326
- [Background] Vazquez B, Shah B, Zhang X, Lash JP, Gordeuk VR, Saraf SL. Hyperfiltration is associated with the development of microalbuminuria in patients with sickle cell anemia. Am J Hematol. 2014 Dec;89(12):1156-7. doi: 10.1002/ajh.23817. Epub 2014 Aug 27. No abstract available. PMID 25132221
- [Background] Ataga KI, Zhou Q, Saraf SL, Hankins JS, Ciccone EJ, Loehr LR, Ashley-Koch AE, Garrett ME, Cai J, Telen MJ, Derebail VK. Longitudinal study of glomerular hyperfiltration in adults with sickle cell anemia: a multicenter pooled analysis. Blood Adv. 2022 Aug 9;6(15):4461-4470. doi: 10.1182/bloodadvances.2022007693. PMID 35696734
- [Background] Aygun B, Mortier NA, Smeltzer MP, Hankins JS, Ware RE. Glomerular hyperfiltration and albuminuria in children with sickle cell anemia. Pediatr Nephrol. 2011 Aug;26(8):1285-90. doi: 10.1007/s00467-011-1857-2. Epub 2011 May 11. PMID 21559933
- [Background] Lebensburger JD, Aban I, Pernell B, Kasztan M, Feig DI, Hilliard LM, Askenazi DJ. Hyperfiltration during early childhood precedes albuminuria in pediatric sickle cell nephropathy. Am J Hematol. 2019 Apr;94(4):417-423. doi: 10.1002/ajh.25390. Epub 2019 Jan 8. PMID 30592084
- [Background] Ware RE, Rees RC, Sarnaik SA, Iyer RV, Alvarez OA, Casella JF, Shulkin BL, Shalaby-Rana E, Strife CF, Miller JH, Lane PA, Wang WC, Miller ST; BABY HUG Investigators. Renal function in infants with sickle cell anemia: baseline data from the BABY HUG trial. J Pediatr. 2010 Jan;156(1):66-70.e1. doi: 10.1016/j.jpeds.2009.06.060. PMID 19880138
- [Background] Amin R, Turner C, van Aken S, Bahu TK, Watts A, Lindsell DR, Dalton RN, Dunger DB. The relationship between microalbuminuria and glomerular filtration rate in young type 1 diabetic subjects: The Oxford Regional Prospective Study. Kidney Int. 2005 Oct;68(4):1740-9. doi: 10.1111/j.1523-1755.2005.00590.x. PMID 16164650
- [Background] Ataga KI, Zhou Q, Derebail VK, Saraf SL, Hankins JS, Loehr LR, Garrett ME, Ashley-Koch AE, Cai J, Telen MJ. Rapid decline in estimated glomerular filtration rate in sickle cell anemia: results of a multicenter pooled analysis. Haematologica. 2021 Jun 1;106(6):1749-1753. doi: 10.3324/haematol.2020.267419. PMID 33179474
- [Background] Niss O, Lane A, Asnani MR, Yee ME, Raj A, Creary S, Fitzhugh C, Bodas P, Saraf SL, Sarnaik S, Devarajan P, Malik P. Progression of albuminuria in patients with sickle cell anemia: a multicenter, longitudinal study. Blood Adv. 2020 Apr 14;4(7):1501-1511. doi: 10.1182/bloodadvances.2019001378. PMID 32289161
- [Background] Alvarez O, Lopez-Mitnik G, Zilleruelo G. Short-term follow-up of patients with sickle cell disease and albuminuria. Pediatr Blood Cancer. 2008 Jun;50(6):1236-9. doi: 10.1002/pbc.21520. PMID 18293385
- [Background] Dharnidharka VR, Dabbagh S, Atiyeh B, Simpson P, Sarnaik S. Prevalence of microalbuminuria in children with sickle cell disease. Pediatr Nephrol. 1998 Aug;12(6):475-8. doi: 10.1007/s004670050491. PMID 9745872
- [Background] Day TG, Drasar ER, Fulford T, Sharpe CC, Thein SL. Association between hemolysis and albuminuria in adults with sickle cell anemia. Haematologica. 2012 Feb;97(2):201-5. doi: 10.3324/haematol.2011.050336. Epub 2011 Oct 11. PMID 21993677
- [Background] Becton LJ, Kalpatthi RV, Rackoff E, Disco D, Orak JK, Jackson SM, Shatat IF. Prevalence and clinical correlates of microalbuminuria in children with sickle cell disease. Pediatr Nephrol. 2010 Aug;25(8):1505-11. doi: 10.1007/s00467-010-1536-8. Epub 2010 May 27. PMID 20505954
- [Background] Saraf SL, Zhang X, Kanias T, Lash JP, Molokie RE, Oza B, Lai C, Rowe JH, Gowhari M, Hassan J, Desimone J, Machado RF, Gladwin MT, Little JA, Gordeuk VR. Haemoglobinuria is associated with chronic kidney disease and its progression in patients with sickle cell anaemia. Br J Haematol. 2014 Mar;164(5):729-39. doi: 10.1111/bjh.12690. Epub 2013 Dec 12. PMID 24329963
- [Background] Ataga KI, Derebail VK, Archer DR. The glomerulopathy of sickle cell disease. Am J Hematol. 2014 Sep;89(9):907-14. doi: 10.1002/ajh.23762. Epub 2014 Jun 19. PMID 24840607
- [Background] Guasch A, Navarrete J, Nass K, Zayas CF. Glomerular involvement in adults with sickle cell hemoglobinopathies: Prevalence and clinical correlates of progressive renal failure. J Am Soc Nephrol. 2006 Aug;17(8):2228-35. doi: 10.1681/ASN.2002010084. Epub 2006 Jul 12. PMID 16837635
- [Background] McClellan AC, Luthi JC, Lynch JR, Soucie JM, Kulkarni R, Guasch A, Huff ED, Gilbertson D, McClellan WM, DeBaun MR. High one year mortality in adults with sickle cell disease and end-stage renal disease. Br J Haematol. 2012 Nov;159(3):360-7. doi: 10.1111/bjh.12024. Epub 2012 Sep 12. PMID 22967259
- [Background] Nissenson AR, Port FK. Outcome of end-stage renal disease in patients with rare causes of renal failure. I. Inherited and metabolic disorders. Q J Med. 1989 Nov;73(271):1055-62. PMID 2516341
- [Background] Powars DR, Elliott-Mills DD, Chan L, Niland J, Hiti AL, Opas LM, Johnson C. Chronic renal failure in sickle cell disease: risk factors, clinical course, and mortality. Ann Intern Med. 1991 Oct 15;115(8):614-20. doi: 10.7326/0003-4819-115-8-614. PMID 1892333
- [Background] Saraf S, Farooqui M, Infusino G, Oza B, Sidhwani S, Gowhari M, Vara S, Gao W, Krauz L, Lavelle D, DeSimone J, Molokie R, Saunthararajah Y. Standard clinical practice underestimates the role and significance of erythropoietin deficiency in sickle cell disease. Br J Haematol. 2011 May;153(3):386-92. doi: 10.1111/j.1365-2141.2010.08479.x. Epub 2011 Mar 21. PMID 21418176
- [Background] Elmariah H, Garrett ME, De Castro LM, Jonassaint JC, Ataga KI, Eckman JR, Ashley-Koch AE, Telen MJ. Factors associated with survival in a contemporary adult sickle cell disease cohort. Am J Hematol. 2014 May;89(5):530-5. doi: 10.1002/ajh.23683. Epub 2014 Feb 21. PMID 24478166
- [Background] Wierenga KJ, Hambleton IR, Lewis NA. Survival estimates for patients with homozygous sickle-cell disease in Jamaica: a clinic-based population study. Lancet. 2001 Mar 3;357(9257):680-3. doi: 10.1016/s0140-6736(00)04132-5. PMID 11247552
- [Background] Gardner K, Douiri A, Drasar E, Allman M, Mwirigi A, Awogbade M, Thein SL. Survival in adults with sickle cell disease in a high-income setting. Blood. 2016 Sep 8;128(10):1436-8. doi: 10.1182/blood-2016-05-716910. Epub 2016 Jul 20. No abstract available. PMID 27439910
- [Background] Darbari DS, Wang Z, Kwak M, Hildesheim M, Nichols J, Allen D, Seamon C, Peters-Lawrence M, Conrey A, Hall MK, Kato GJ, Taylor JG 6th. Severe painful vaso-occlusive crises and mortality in a contemporary adult sickle cell anemia cohort study. PLoS One. 2013 Nov 5;8(11):e79923. doi: 10.1371/journal.pone.0079923. eCollection 2013. PMID 24224021
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Powars DR, Chan LS, Hiti A, Ramicone E, Johnson C. Outcome of sickle cell anemia: a 4-decade observational study of 1056 patients. Medicine (Baltimore). 2005 Nov;84(6):363-376. doi: 10.1097/01.md.0000189089.45003.52. PMID 16267411
- [Background] Quinn CT, Rogers ZR, McCavit TL, Buchanan GR. Improved survival of children and adolescents with sickle cell disease. Blood. 2010 Apr 29;115(17):3447-52. doi: 10.1182/blood-2009-07-233700. Epub 2010 Mar 1. PMID 20194891